CLINICAL TRIAL: NCT00404313
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter, Parallel-Group, Dose-Ranging Study of MK0633 in Adult Patients With Chronic Asthma
Brief Title: The Effect of MK0633 in Patients With Chronic Asthma (0633-007)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0633-007; MK0633-007; 2006_553
Record Dates: First submitted 2006-11-21; First posted 2006-11-28 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — MK-0633 p-toluenesulfonate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): MK0633 10 mg
  Interventions: Drug: MK0633
- 2 (Experimental): MK0633 50 mg
  Interventions: Drug: MK0633
- 3 (Experimental): MK0633 100 mg
  Interventions: Drug: MK0633
- 4 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: MK0633 — Patients will receive 10 mg, 50 mg, or 100 mg MK0633 tablets once daily for 6 weeks. There will be 2 week period during which all patients will receive placebo to MK0633
  Arms: 1; 2; 3
Drug: Comparator: placebo — Placebo to MK0633 10 mg, 50 mg, or 100 mg tablets once daily for 6 weeks
  Arms: 4

SUMMARY:
A clinical study to evaluate the efficacy and safety of MK0633 in adult patients with chronic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical history of symptoms of chronic asthma, including dyspnea, wheezing, chest tightness, cough, and/or sputum production
* Males and females 18-70 years of age

Exclusion Criteria:

* History of kidney or chronic liver disease
* Recent history of heart problems within the past 3 months
* Evidence of another clinically significant, active lung disorder such as bronchiectasis or COPD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test data measured over 6 weeks | 6 weeks

SECONDARY OUTCOMES:
Overall daytime and nighttime symptoms score, beta-agonist use, asthma exacerbations, asthma-specific quality of life questionnaire score, measured over 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Wasfi YS, Villaran C, de Tilleghem Cle B, Smugar SS, Hanley WD, Reiss TF, Knorr BA. The efficacy and tolerability of MK-0633, a 5-lipoxygenase inhibitor, in chronic asthma. Respir Med. 2012 Jan;106(1):34-46. doi: 10.1016/j.rmed.2011.08.019. Epub 2011 Sep 25. PMID 21945511